CLINICAL TRIAL: NCT04445701
Title: A Phase 1/2, Dose Escalation Safety and Tolerability Study of AO-176 as Monotherapy and in Combination With Bortezomib and Dexamethasone in Adults With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of AO-176 as Monotherapy and in Combination With Bortezomib/Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arch Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AO-176-102
Record Dates: First submitted 2020-06-17; First posted 2020-06-24 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: AO-176; CD47; Immunotherapy; Monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase 1 Part 1: Up to 4 dose escalation cohorts will be enrolled; each cohort will initially recruit 3 patients to receive AO-176 monotherapy in a standard 3+3 design; the cohort will be expanded in the event of a DLT. Once the RP2D has been identified, an expansion cohort will be enrolled to evaluate AO-176 at the RP2D in combination with dexamethasone (DEX).
  Phase 1 Part 2: Dose escalation cohorts will evaluate AO-176 in combination with DEX and bortezomib (BORT) to determine the RP2D of AO-176 + DEX + BORT in a standard 3+3 design; the cohort will be expanded in the event of a DLT.
  Phase 2: Up to 48 patients will be enrolled to evaluate the preliminary efficacy of AO-176 + DEX + BORT using a Simon 2-stage design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AO-176 Dose Escalation Monotherapy (Experimental): The dose escalation monotherapy cohorts will initially recruit 3 patients to receive AO-176 in a standard 3+3 design; cohorts will be expanded in the event of a DLT.
  Interventions: Drug: AO-176
- AO-176 + DEX Expansion Cohort (Experimental): Once the monotherapy RP2D has been established, an expansion cohort of AO-176 + dexamethasone will be enrolled.
  Interventions: Drug: AO-176 + Dex
- AO-176 + DEX + BORT Dose Escalation (Experimental): Following evaluation of AO-176 + dexamethasone, dose escalation cohorts of AO-176 + dexamethasone + bortezomib will be enrolled. Each dose escalation cohort will initially recruit 3 patients in a standard 3+3 design; cohorts will be expanded in the event of a DLT. The Phase 2 portion of the study will further evaluate the RP2D of AO-176 + DEX + BORT.
  Interventions: Drug: AO-176 + Dex + Bort

INTERVENTIONS:
Drug: AO-176 — Humanized monoclonal antibody (mAb) targeting CD47
  Arms: AO-176 Dose Escalation Monotherapy
Drug: AO-176 + Dex — Humanized mAb targeting CD47 plus dexamethasone
  Arms: AO-176 + DEX Expansion Cohort
Drug: AO-176 + Dex + Bort — Humanized mAb targeting CD47 plus dexamethasone plus bortezomib
  Arms: AO-176 + DEX + BORT Dose Escalation

SUMMARY:
Open-label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics (PK)/pharmacodynamics and initial efficacy of AO-176 as monotherapy and in combination with dexamethasone and bortezomib in adults with relapsed/refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
An open-label, multicenter, dose escalation study to evaluate the safety, tolerability and PK/pharmacodynamics of AO-176 in adults with relapsed/refractory multiple myeloma whose disease has progressed following at least 3 prior systemic lines of treatment and must have progressed on the final line of therapy received before being considered for this study.

The study will be conducted in 2 phases; Phase 1 is an ascending-dose study of AO-176 monotherapy utilizing the classic 3+3 design, with enrollment of 3 patients per cohort and expansion of the cohort in the event of a dose-limiting toxicity (DLT). Following the dose escalation portion and determination of the monotherapy recommended phase 2 dose (RP2D), an ascending dose escalation study of AO-176 and dexamethasone combined with bortezomib will be evaluated utilizing the same 3+3 dose escalation design.

Phase 2 will evaluate the clinical activity of AO-176 plus dexamethasone and bortezomib at the RP2D as determined in Phase 1 Part 2.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of symptomatic MM per IMWG criteria
2. Measurable disease
3. Relapsed or refractory to at least 3 prior systemic lines of therapy for MM
4. Eastern Cooperative Oncology Group (ECOG) status 0-2
5. Resolution of prior therapy-related adverse events
6. Minimum of 2 weeks since last dose of cancer therapy or radiotherapy

Key Exclusion Criteria:

1. Previous Grade 3-4 infusion or hypersensitivity reaction
2. Severe asthma or chronic obstructive pulmonary disease exacerbations requiring hospital admission or steroids
3. Prior treatment with a checkpoint inhibitor (anti-PD-1, PD-L1 or CTLA-4) within 4 weeks.
4. Prior treatment with a therapeutic agent that targets the CD47 axis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Phase 1: MTD / RP2D of AO-176 assessed by incidence of dose-limiting toxicities and incidence of treatment-related adverse events (TEAEs) as assessed by CTCAE v5.0 | 12 months
  Safety and tolerability of AO-176 when administered as monotherapy and in combination with dexamethasone or with dexamethasone plus bortezomib in adult patients with R/R MM as assessed by incidence of DLTs and TEAEs as assessed by CTCAE v5.0
Phase 2: Objective response rate (ORR) of AO-176 + DEX + BORT | 12 months
  Evaluate the clinical activity of AO-176 + dexamethasone + bortezomib based on ORR using International Myeloma Working Group (IMWG) uniform response criteria

SECONDARY OUTCOMES:
Phase 1: ORR of single agent AO-176 | 12 months
  Evaluate the clinical activity of single agent AO-176 based on ORR using IMWG uniform response criteria
Phase 1: Duration of response (DOR) of single agent AO-176 | 12 months
  Evaluate the clinical activity of single agent AO-176 based on DOR using IMWG uniform response criteria
Phase 1: Disease control rate (DCR) of single agent AO-176 | 12 months
  Evaluate the clinical activity of single agent AO-176 based on DCR using IMWG uniform response criteria
Phase 1: Progression-free survival (PFS) of single agent AO-176 | 12 months
  Evaluate the clinical activity of single agent AO-176 based on PFS using IMWG uniform response criteria
Phase 1: Overall survival (OS) of single agent AO-176 | 12 months
  Evaluate the clinical activity of single agent AO-176 based on OS
Phase 2: DOR of AO-176 + DEX + BORT | 12 months
  Evaluate the clinical activity of AO-176 + dexamethasone + bortezomib based on DOR using IMWG uniform response criteria
Phase 2: DCR of AO-176 + DEX + BORT | 12 months
  Evaluate the clinical activity of AO-176 + dexamethasone + bortezomib based on DCR using IMWG uniform response criteria
Phase 2: PFS of AO-176 + DEX + BORT | 12 months
  Evaluate the clinical activity of AO-176 + dexamethasone + bortezomib based on PFS using IMWG uniform response criteria
Phase 2: OS of AO-176 + DEX + BORT | 12 months
  Evaluate the clinical activity of AO-176 + dexamethasone + bortezomib based on OS

CONTACTS AND LOCATIONS:
Overall Officials: Ben Oshrine, MD, Study Director — Sr Medical Director, Arch Oncology
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrejeva G, Capoccia BJ, Hiebsch RR, Donio MJ, Darwech IM, Puro RJ, Pereira DS. Novel SIRPalpha Antibodies That Induce Single-Agent Phagocytosis of Tumor Cells while Preserving T Cells. J Immunol. 2021 Feb 15;206(4):712-721. doi: 10.4049/jimmunol.2001019. Epub 2021 Jan 11. PMID 33431660